CLINICAL TRIAL: NCT05243121
Title: Peking University People's Hospital Radiology
Brief Title: Artificial Intelligence Analysis for Magnetic Resonance Imaging in Screening and Diagnosis of Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, WangYi, Director, Peking University People's Hospital
Other Study IDs: AI-BMRI-S
Record Dates: First submitted 2021-09-12; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Breast Neoplasms; Magnetic Resonance Imaging
Keywords: breast neoplasms; magnetic resonance imaging; screening; deep learning; machine learning
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinically symptomatic patients: Clinically symptomatic patients (defined as palpable masses, nipple discharge, asymmetric thickening or nodules, and abnormal skin changes according to the guidelines) should be examined by BMRI at the judgment of the clinician.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — undergoing enhanced MRI

SUMMARY:
Use Convolutional Neural Networks Analysis for Classification of Contrast-enhancing Lesions at Multiparametric Breast MRI. Build an abbreviated protocal, and investigate whether an abbreviated protocol was suitable for breast magnetic resonance imaging screening for breast mass in Chinese women, which can shorten the examination time and avoid enhanced imaging while ensuring the accuracy of the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical symptoms (define as palpable mass, nipple discharge, asymmetric thickening or nodules, and abnormal skin changes)
* Patients undergoing full sequence BMRI examination
* Through the follow-up database, at least 6 months of follow-up results can be obtained to determine whether the diagnosis result is negative/benign/malignant; for patients who need pathological biopsy, the pathological biopsy results shall prevail to determine the lesion benign/malignant

Exclusion Criteria:

* The breast had received radiotherapy, chemotherapy, biology and other treatments before BMRI.
* There are contraindications for breast-enhanced MRI examinations such as allergy to contrast agents.
* A prosthesis is implanted in the affected breast.
* Patients during lactation or pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Study Population: Clinically symptomatic patients (defined as palpable masses, nipple discharge, asymmetric thickening or nodules, and abnormal skin changes according to the guidelines) should be examined by BMRI at the judgment of the clinician.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Breast Cancer Screening | 5 years
  Compare the area under the curve of the deep learning model of the BMRI full sequence, contrast-enhanced and non-contrast-enhanced sequence in the diagnosis of breast cancer.

SECONDARY OUTCOMES:
The accuracy of radiologists and deep learning models | 5 years
  Under the conditions of BMRI full sequence, contrast-enhanced and non-contrast-enhanced sequences, compare the sensitivity, specificity, positive predictive value and negative predictive value of breast tumor detection by radiologists and deep learning models.
Health economics | 5 years
  Compare the examination time, reading time and cost of BMRI full sequence, contrast-enhanced and non-contrast-enhanced sequences.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university people's hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No